CLINICAL TRIAL: NCT00990613
Title: A Phase 1, Fixed Sequence, Cross-Over Study To Investigate The Single Dose Pharmacokinetics Of A Dimebon (Latrepirdine) Transdermal Solution Relative To The Immediate Release Formulation In Older Adults
Brief Title: A Study Evaluating The Absorption Of Dimebon Into The Body From A Dimebon Solution Applied To The Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: B1451038
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Alzheimer's Disease; Huntington's Disease
Keywords: percutaneous transcutaneous dimebon transdermal pharmacokinetics
MeSH Terms: conditions — Alzheimer Disease; Huntington Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Other)
  Interventions: Drug: Dimebon IR; Drug: Dimebon Transdermal
- Cohort 2 (Other)
  Interventions: Drug: Dimebon IR; Drug: Dimebon Transdermal

INTERVENTIONS:
Drug: Dimebon IR — A single, oral 10 mg dose of dimebon dihydrochloride (equivalent to 8.2 mg free base) immediate release will be administered.
  Arms: Cohort 1
Drug: Dimebon Transdermal — A single, transdermal 5 mg dose of dimebon free base solution will be applied to the back over a 24 hour period. A double-blinded vehicle (placebo) solution will be applied concurrently to a contralateral body site.
  Arms: Cohort 1
Drug: Dimebon Transdermal — A single, to be determined dose of dimebon free base solution will be applied to the back over a 24 hour period. The dose level chosen will be determined based on the pharmacokinetic/safety profile of the 5 mg dose. A double-blinded vehicle (placebo) solution will be applied concurrently to a contralateral body site.
  Arms: Cohort 1
Drug: Dimebon IR — A single, oral 10 mg dose of dimebon dihydrochloride (equivalent to 8.2 mg free base) immediate release will be administered.
  Arms: Cohort 2
Drug: Dimebon Transdermal — A single, to be determined dose of dimebon free base solution will be applied to the back over a 24 hour period. The dose level chosen will be determined based on the pharmacokinetic/safety profile of the 5 mg dose in Cohort 1. A double-blinded vehicle (placebo) solution will be applied concurrently to a contralateral body site.
  Arms: Cohort 2

SUMMARY:
To estimate the absorption, safety, and tolerability of a dimebon transdermal solution relative to the dimebon immediate release oral formulation.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian, male or females, 50 to 85 years inclusive.
* Subjects must have adequate space available on each side of the upper or middle back that is free from excessive hair, broken or irritated skin, tattoos, scars, moles, acne, and sunburn.

Exclusion Criteria:

* Evidence or history of any major medical or psychiatric illness or unstable medical condition within six months of Screening that may increase the risk associated with study participation.
* Subjects with any central nervous system disease including Alzheimer's disease, Parkinson's disease, Huntington disease, or any form of dementia.
* Subjects with any history of stroke, known cerebrovascular disease or subjects with any history of structural brain disease.
* Any history of epilepsy, seizure disorder (i.e., including febrile seizures) or convulsion.
* Subjects with any skin disorders that might prevent application of the dimebon solution including, but not limited to, any known sensitivity to adhesives.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic endpoints include dimebon area under the curve from 0 to the last quantifiable concentration (AUClast) and dimebon area under the curve from 0 to infinity (AUCinf) as permitted by data | 4 to 6 days

SECONDARY OUTCOMES:
Safety endpoints include subjective symptoms/objective findings (including skin irritation), clinical safety laboratory assessments, 12 lead ECGs, and supine vital signs. | 4 to 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Kalamazoo, Michigan, United States

REFERENCES:
- [Derived] Chew ML, Mordenti J, Yeoh T, Ranade G, Qiu R, Fang J, Liang Y, Corrigan B. Minimization of CYP2D6 Polymorphic Differences and Improved Bioavailability via Transdermal Administration: Latrepirdine Example. Pharm Res. 2016 Aug;33(8):1873-80. doi: 10.1007/s11095-016-1922-4. Epub 2016 Apr 12. PMID 27072954
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1451038&StudyName=A%20Study%20Evaluating%20The%20Absorption%20Of%20Dimebon%20Into%20The%20Body%20From%20A%20Dimebon%20Solution%20Applied%20To%20The%20Skin